CLINICAL TRIAL: NCT01763073
Title: Beliefs and Practice Intentions of Future Ob/Gyn Residents Regarding Reproductive Healthcare
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Principal Investigator, Instructor, Brigham and Women's Hospital
Other Study IDs: 2012P001794
Record Dates: First submitted 2013-01-03; First posted 2013-01-08 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Focus: Pre-residency Intention to Provide Abortion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medical Students: Fourth-year students in accredited US medical schools who have applied to, but not yet been matched with, residency programs in obstetrics and gynecology.

SUMMARY:
The objective of this study is to ascertain factors shaping medical students' pre-residency intention to provide abortion through an in-depth qualitative investigation into the context and experiences that shape intention to provide.

ELIGIBILITY:
Inclusion Criteria:

* current 4th-year medical student
* US accredited medical school
* has applied to, but not yet been accepted into, obstetrics and gynecology residency programs

Exclusion Criteria:

* age less than 18 years
* former student reapplying to residency (e.g., not current 4th-year student)
* has not yet applied to residency
* has already been accepted to residency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fourth-year students in accredited US medical schools who have applied to, but not yet been matched with, residency programs in obstetrics and gynecology.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Factors affecting pre-residency intention to provide abortion | Up to 15 months. Each participant will be interviewed once, between January and March 2013 or between September 2013 through March 2014.
  Factors will be identified by systematically coding qualitative data using a combination of deductive and inductive analytical strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States